CLINICAL TRIAL: NCT06787716
Title: Impact of Whole-body Vibration Training on Flexibility, Muscular Activity and Quality of Life After Lower Extremity Thermal Burn Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rokaia Ali Zainelabedeen Mohamed Toson, Assistant Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005595
Record Dates: First submitted 2024-12-26; First posted 2025-01-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Lower Extremity Burns
Keywords: burn; flexibility; EMG; muscular activity; quality of life
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole body vibration group (Experimental)
  Interventions: Device: The whole body vibration
- Control group (Other)
  Interventions: Other: The traditional physical therapy program

INTERVENTIONS:
Device: The whole body vibration — Patients in the study group will receive the traditional physical therapy program first (passive and active ROM exercises, stretching and strengthening exercises) for 60 minutes, 3 days/ week for 12 weeks.This will be followed immediately by whole-body vibration training on the vibration platform (Power Plate International, Irvine, California, USA) at the same visit. The vibration frequency will be 30 Hz and the amplitude from 4 to 7 mm, with an increase of 1mm every two weeks. The WBV program will be three sessions a week for 12 weeks. WBV duration started with 10 min at the 1st week up to 35 min at the 12th week, with a regular increase of five minutes every two successive weeks.
  Arms: Whole body vibration group
Other: The traditional physical therapy program — The traditional physical therapy program will be three days a week for 12 weeks. The program will include 60 minutes of a supervised and individualized exercise program including passive and active exercises of the hip, knee, and ankle joints, stretching exercises for the Calf and hamstring muscles followed by strengthening exercises of the hip, knee, ankle, and foot muscles. To improve the strength, free weights will be used for all exercises. During the first week, 50 to 60% of the repetitions maximum test will be set as the starting weight. Then, from the second week to the sixth, the weight will be increased to 70%-75% of three repetitions maximum (3 sets, 4-10 repetitions). The training amplitude then will be raised to 80%-85% of the three-repetition maximum (3 sets, 8-12 repetitions) that will be continued through weeks 7 to 12, holding 5 seconds at the end of the range.
  Arms: Control group

SUMMARY:
Tight hamstring muscles limit the anterior tilt of the pelvis in spinal flexion resulting in aggravated muscle and ligamentous tension in the lumbar region which leads to significantly higher compressive loads on the lumbar spine. Other postural changes associated with tightness of the hamstrings can influence the sacroiliac joint stability in an indirect way. Hence, flexibility of hamstring muscles is crucial for overall well-being and optimal physical fitness.

ELIGIBILITY:
Inclusion criteria:

1. Patients with a deep second-degree thermal burn of the lower extremity, 35%-40% total body surface area (TBSA) of burn as measured with the rule of nine, after six weeks from the injury or complete wound healing.
2. Patients with 20 to 50 years old.
3. Absence of any neurological disorder i.e.: stroke, ataxia, or parkinsonism.

Exclusion criteria:

1. Patients with open wounds.
2. Patients with recent fractures.
3. Patients with severe obesity BMI ≥40.
4. Patients with cardiorespiratory disorders.
5. Patients with bone disease, joint replacement, and traumatic spine history since last year.

In order to apply the inclusion and exclusion criteria, all cases will be subjected to an interview and assessment.

Those subjects who will be eligible to take part in the study will sign an informed consent before participation in the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test: | 12 weeks
  Active knee extension test: The knee extension angle was measured using a standard goniometer. The goniometer was placed at the lateral epicondyle of the femur, with one arm aligned with the femur and the other with the tibia.

SECONDARY OUTCOMES:
Straight Leg Raising Test | 12 weeks
  The straight leg raising test will be used to determine the hip flexion angle by using a standard goniometer. The fixed arm will be parallel to the table, while the other will point to the lateral femoral condyle and malleolus. At the point of discomfort, the goniometer will be oriented with the movable arm toward the lateral malleolus.
Electromyography for Quadriceps Muscle | 12 weeks
  Electromyography will be used to assess the activity of the following muscles at baseline then at the end of the 12 weeks intervention: Vastus medialis, vastus lateralis and rectus femoris.
Electromyography for Hamstring Muscles | 12 weeks
  Electromyography will be used to assess the activity of the following muscles at baseline then at the end of the 12 weeks intervention: Biceps femoris and medial hamstrings.
The SF-36 questionnaire | 6 months
  SF-36 is a health related quality of life measure with 35 of the items related to one of the 8 health concepts. One item addresses health transition and is not included in the scoring. The health concepts measured include physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.
  The SF-36 Subscales (Each scored 0-100)
  * Physical Functioning (PF)
  * Role Limitations - Physical (RP)
  * Bodily Pain (BP)
  * General Health (GH)
  * Vitality (VT)
  * Social Functioning (SF)
  * Role Limitations - Emotional (RE)
  * Mental Health (MH)
  Interpretation:
  0 = Worst possible health status for that domain 100 = Best possible health status for that domain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Giza Governorate, Egypt